CLINICAL TRIAL: NCT03040934
Title: A Prospective, Open Label, Multi-center Trial of Firehawk™ Coronary Stent System in the Treatment of Coronary Chronic Total Occlusion Lesion(s) by Optical Coherent Tomography (OCT) and Coronary Angiography
Brief Title: Firehawk™ Coronary Stent System in the Treatment of Coronary Chronic Total Occlusion Lesion(s)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGET CTO
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Drug-Eluting Stents; Percutaneous Coronary Intervention; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firehawk implantation (Active Comparator): 98 subjects will be enrolled to receive a test device (Firehawk™).
  Interventions: Device: Firehawk sirolimus target eluting coronary stent system
- XIENCE implantation (Active Comparator): 98 subjects will be enrolled to receive a control device (XIENCE).
  Interventions: Device: XIENCE Everolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Firehawk sirolimus target eluting coronary stent system — 98 subjects will be enrolled to receive a test device of Firehawk sirolimus target eluting coronary stent system
  Other Names: Firehawk™
  Arms: Firehawk implantation
Device: XIENCE Everolimus-Eluting Coronary Stent System — 98 subjects will be enrolled to receive a control device of XIENCE Everolimus-Eluting Coronary Stent System
  Other Names: XIENCE EES
  Arms: XIENCE implantation

SUMMARY:
This study is a prospective, multi-center, open-label, randomized controlled clinical trial,aims to assess the safety and effectiveness of the Firehawk™ sirolimus target-eluting coronary stent system with abluminal grooves containing a biodegradable polymer (Firehawk™) comparing the XIENCE everolimus-eluting coronary stent system in the treatment of subjects with total coronary occlusion lesion(s).

DETAILED DESCRIPTION:
This study will recruit 196 subjects with total coronary occlusion lesion(s) in coronary arteries ≥2.25 mm to ≤4.0 mm in diameter and ≤100 mm in length (by visual estimate) in no more than 10 research centers in China. All participants met the inclusion criteria will be 1:1 randomized to receive Firehawk™ sirolimus target-eluting coronary stent or XIENCE everolimus-eluting coronary stent.

Optical Coherent Tomography (OCT) sub study: the first 44 consecutive subjects who consented to participate in the OCT sub study will undergo OCT assessment at 3 months and 12 months post index procedure. The OCT sub study will be performed in 3-5 pre-selected sites. The clinical follow-up will be carried out at 30 days, 3 months, 6 months, 12 months,and 2-5 years post-index procedure.The primary endpoint is in-stent late lumen loss at 12 months post-index procedure.The secondary endpoint is neo-intimal thickness by Optical Coherent Tomography (OCT) at 3 months post-index procedure.

ELIGIBILITY:
Clinical Inclusion Criteria:

* CI1. Subject must be at least 18 years of age;
* CI2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;
* CI3. Subject is eligible for percutaneous coronary intervention (PCI);
* CI4. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia;
* CI5. Subjects are eligible candidates for coronary artery bypass graft surgery (CABG);
* CI6. Left ventricular ejection fraction (LVEF) within 60 days ≥ 35%; Exclusion Criteria;
* CI7. Subject is willing to comply with all protocol-required follow-up evaluation.

Angiographic Inclusion Criteria (visual estimate):

* AI1. Target lesions must be new and have a visually estimated reference diameter ≥2.25 mm and ≤4.0 mm in autologous coronary artery;
* AI2. Target lesions must be < 100 mm in length (visual estimate) and the number of implanted stents is less than 4;
* AI3. Target lesions must be visually complete occlusion and longer than 4 weeks;
* AI4. Target lesions must be able to pass and be successfully expanded;

Clinical Exclusion Criteria:

* CE1. Subjects recently suffer from MI (within 1 week), and ECG changes/clinical symptoms consistent with AMI or accompanied with increased cardiac biomarkers (CK-MB, CK, TNT or TNI) are excluded;
* CE2. Subjects had an organ transplant or are waiting for an organ transplant;
* CE3. Subjects are receiving chemotherapy or will receive a chemotherapy within 30 days after PCI;
* CE4. Subjects are undergoing chronic (over 72 hours) anticoagulant therapy (such as heparin and coumarin) other than acute coronary syndrome;
* CE5. Subjects with abnormal counts of platelet and white blood cell (WBC): platelet counts less than 100×10E9/L or greater than 700×10E9/L, white blood cells less than 3×10E9/L;
* CE6. Subjects have confirmed or suspected liver disease, including hepatitis lab results;
* CE7. Subjects with elevated serum creatinine level >3.0mg/dL or undergoing dialysis therapy;
* CE8. Subjects with active peptic ulcer, active gastrointestinal (GI) bleeding or other bleeding diathesis or coagulopathy, or refused a blood transfusion;
* CE9. Subjects with cerebral vascular accident (CVA) or transient ischemic attack (TIA) in the past 6 months, or with permanent nerve defects;
* CE10. Subjects had any PCI (such as balloon angioplasty, stent, cutting balloon,atherectomy) treatment in target vessels (including collateral) within 12 months prior to baseline;
* CE11. Subjects plan to undergo PCI or CABG after the baseline PCI;
* CE12. Subjects have any coronary endovascular brachytherapy treatment previously;
* CE13. Subjects associated with drugs allergy (such as sirolimus, or structure-related compounds fluorinated polymers, thiophenepyridine or aspirin);
* CE14. Subjects are suffering from other serious illness (such as cancer, congestive heart failure), which may cause drop in life expectancy to less than 18 months;
* CE15. Subjects are currently abusing drugs (such as alcohol, cocaine, heroin, etc);
* CE16. Subject plan to undergo any operations that may lead to confuse with the programme;
* CE17. Subjects were participating in another study of drug or medical device which did not meet its primary endpoint;
* CE18. Subjects plan to pregnant within 18 months after baseline;
* CE19. Subjects are pregnant or breastfeeding women.

Angiographic Exclusion Criteria (visual estimate):

* AE1. Target lesions with the following criteria: left main, saphenous vein grafts or arterial grafts, via saphenous vein grafts or arterial graft, and in-stent stenosis;
* AE2. Subjects with unprotected left main coronary artery disease (diameter stenosis >50%);
* AE3. Subjects have a protected left main coronary artery disease (diameter stenosis> 50% and left coronary artery bypass surgery), as well as target lesions located in the LAD and LCX;
* AE4. Subjects with other lesions of clinical significance, may be need intervention within 18 months after baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
In-stent late lumen loss | At 12 months post-index procedure

SECONDARY OUTCOMES:
Neo-intimal thickness by Optical Coherence Tomography (OCT) | At 3 months post-index procedure

OTHER OUTCOMES:
Target Vessel Failure (TVF) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Target Lesion Failure (TLF) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Target Vessel Revascularization (TVR) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Target Lesion Revascularization (TLR) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Myocardial Infarction (MI,including Q-wave MI and non Q-wave MI) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Death (All cause, Cardiac, Non-cardiac) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Cardiac Death/ All Myocardial Infarction | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
Stent Thrombosis (per ARC definition) | During hospitalization and 30 days, 3 months, 6 months, 12 months and 2-5 years post-index procedure.
In-stent and in-segment percent diameter stenosis (DS%) | At 12 months post-index procedure.
In-segment late lumen loss | At 12 months post-index procedure.
In-stent and in-segment minimum lumen diameter (MLD) | At 12 months post-index procedure.
In-stent and in-segment binary restenosis rate (%) | At 12 months post-index procedure.
Mean/Minimal Stent area (mm2) | At 3 months and 12 months post-index procedure.
Mean/Minimal Lumen area (mm2) | At 3 months and 12 months post-index procedure.
Lumen volume (mm3) | At 3 months and 12 months post-index procedure.
Stent volume (mm3) | At 3 months and 12 months post-index procedure.
Mean neointimal hyperplasia area (mm2) | At 3 months and 12 months post-index procedure.
In-stent neointimal hyperplasia volume obstruction (%) | At 3 months and 12 months post-index procedure.
Uncovered strut rate (%) | At 3 months and 12 months post-index procedure.
Malapposed strut rate (%) | At 3 months and 12 months post-index procedure.
Malposed and uncovered strut rate (%) | At 3 months and 12 months post-index procedure.
Technical success rate | Instantly after index procedure.
Clinical procedural success rate | At time of procedure up to 7 days in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Shenyang Military
Locations (1):
- The General Hospital of Shenyang Military, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared. Additionally, study protocol will be available. The data will become available for the beginning 3 months and ending 5 years following article publication. The access criteria are as follow:
  (With) Researchers who provide a methodologically sound proposal. (For the analysis) to achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).
  If the data sharing plan changes after registration, this should be reflected in the statement submitted and published with the manuscript, and updated in the registry record.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: (With) Researchers who provide a methodologically sound proposal. (For the analysis) to achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Derived] Wang G, Zhang R, Chen SL, Wang J, Li Y, Zheng M, Cao R, Ma Y, Sun Z, Li X, Su X, Lu W, Xu Y, Li X, Li Y, Sun F, Han Y; TARGET CTO Investigators. Targeted therapy with a localized abluminal groove low-dose sirolimus-eluting bioabsorbable polymer coronary stent in chronic total occlusions: The TARGET CTO non-inferiority randomized trial. Am Heart J. 2025 Jul;285:93-104. doi: 10.1016/j.ahj.2025.01.018. Epub 2025 Feb 3. PMID 39909342
- [Derived] Wang G, Li Y, Lu W, Xu Y, Su X, Chen S, Li Y, Han Y; TARGET CTO OCT substudy Investigators. Vascular Healing After Biodegradable Polymer Sirolimus-Eluting Versus Durable Polymer Everolimus-Eluting Stents in Chronic Total Occlusions. Catheter Cardiovasc Interv. 2025 Apr;105(5):1124-1133. doi: 10.1002/ccd.31423. Epub 2025 Jan 29. PMID 39878429